CLINICAL TRIAL: NCT03707925
Title: Bronchoscopic Laser Ablation of Solid Peripheral Lung Tumors Followed by Surgical Resection (BLAST-SR Trial)
Brief Title: Bronchoscopic Laser Ablation of Peripheral Lung Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very slow accrual rate
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0474; NCI-2018-02133 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0474 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Lung Carcinoid Tumor; Lung Non-Small Cell Carcinoma; Metastatic Lung Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (bronchoscopic laser ablation, CBCT) (Experimental): Patients undergo bronchoscopic laser ablation following standard bronchoscopy and endobronchial ultrasound. Patients also undergo CBCT before and after laser ablation. 48-72 hours after the procedure, patients undergo standard surgical resection of the lung tumor.
  Interventions: Procedure: Cone-Beam Computed Tomography; Procedure: Conventional Surgery; Procedure: Laser Ablation

INTERVENTIONS:
Procedure: Cone-Beam Computed Tomography — Undergo CBCT
  Other Names: Cone Beam CT
Procedure: Conventional Surgery — Undergo standard resection
Procedure: Laser Ablation — Undergo bronchoscopic laser ablation
  Other Names: ABLATION, LASER; Photoablation

SUMMARY:
As our population ages and we diagnose early lung cancer in patients who cannot undergo surgery due to multiple medical conditions, there is growing interest in minimally invasive modalities to treat these tumors. In this study we are assessing the ability of bronchoscopic laser ablation to kill the cancer cells in these tumors. Patients will undergo bronchoscopy (a tube-like instrument inserted through the mouth to view the inside of the trachea, air passages, and lungs). A thin catheter will be passed through the wind-pipes and into the lung tumor with computed tomography guidance. A laser probe is then passed through this catheter and it is used to destroy the tumor with heat. Patients will then undergo lung surgery with resection of the tumor, and the resected specimen will be reviewed to describe the amount of tumor-kill produced by the laser.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the pathologic changes that result from bronchoscopic laser ablation of peripheral lung tumors focusing on the proportion of complete tumor ablation.

SECONDARY OBJECTIVES:

I. To assess the safety of this technique by describing both procedure-related complications such as bleeding or pneumothorax and post-procedure adverse effects such as fever or pneumonitis.

II. To assess the pathologic changes observed in the lung tissue surrounding the treated lung tumor.

III. To assess radiographic changes observed by cone-beam computed tomography (CT) immediately after the application of bronchoscopic laser ablation.

OUTLINE:

Patients undergo bronchoscopic laser ablation following standard bronchoscopy and endobronchial ultrasound. Patients also undergo CBCT before and after laser ablation. 48-72 hours after the procedure, patients undergo standard surgical resection of the lung tumor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Performance status 0-2 (Eastern Cooperative Oncology Group classification)
* Subject is considered a candidate for bronchoscopy
* Subject is considered a candidate for surgery (other lobar or sub-lobar resection) based on radiographic staging and functional evaluation
* Lung lesion that is either biopsy-proven cancer or is suspicious for cancer
* Both non-small cell lung cancer (including carcinoid tumors) and metastatic disease
* The lesions should be: =< 3 cm, located in the outer 2/3 of the lung, and leave >= 1 cm of tumor-free lung parenchyma between target tumor and pleura or fissure

Exclusion Criteria:

* Tumors greater than 3 cm, located in the inner 1/3 of the lung, invading a major vessel, or located < 1 cm from the pleural or fissure
* Tumors qualified as non-resectable
* Tumors that cannot be reached bronchoscopically
* Patients declared non-surgical candidates
* Patients who are not candidates for bronchoscopy
* Patients with lung cancer who are found to have N2-3 disease
* Patient with lung metastases who are found to have any malignant mediastinal lymph node
* Patients in which the target lesion is confirmed as benign or small cell lung cancer
* Patients without a prior diagnosis of the target lesion whose diagnosis cannot be made during bronchoscopy
* Patients who have received chemotherapy within 60 days prior to bronchoscopic laser ablation
* Patients who were previously treated for the target lesion
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F Casal, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Department of Gynecologic Oncology and Reproductive Medicine at The University of Texas MD Anderson Cancer Center and the Gynecologic Oncology Clinics in the Regional Care Centers.
Pre-assignment Details: 4 participants consented, 1 inevaluable
Groups:
- Bronchoscopic Laser Ablation, Cone-beam CT(CBCT): Patients undergo bronchoscopic laser ablation following standard bronchoscopy and endobronchial ultrasound. Patients also undergo CBCT before and after laser ablation. 48-72 hours after the procedure, patients undergo standard surgical resection of the lung tumor.
  Cone-Beam Computed Tomography: Undergo CBCT
  Conventional Surgery: Undergo standard resection
  Laser Ablation: Undergo bronchoscopic laser ablation
Period: Overall Study
Arm/Group | Bronchoscopic Laser Ablation, Cone-beam CT(CBCT)
Started | 4
Completed | 3
Not Completed | 1
Not completed — Inevaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bronchoscopic Laser Ablation, Cone-beam CT(CBCT)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Changes From Bronchoscopic Laser Ablation of Peripheral Lung Tumors
Description: Pathologic changes will be categorized into three groups: 1. Complete Ablation: absence of staining (anti-mitochondria antibody [MAB] 1273 or nicotinamide adenine dinucleotide-hydrogen [NADH], or both) of tumor cells. 2. Quasi-Complete Ablation: positive staining of 10% of tumor cells. 3. Incomplete ablation: positive staining in > 10% of tumor cells. Will conduct extensive descriptive analyses of the data collected. Will calculate the appropriate summary statistics and 90% confidence intervals (CIs) for the measures of interest.
Time Frame: Up to 16 months
Population: Only patients who underwent bronchoscopic tumor ablation are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Bronchoscopic Laser Ablation, Cone-beam CT(CBCT)
Number analyzed (Participants) | 3
Participants
  Complete Ablation | 0
  Quasi-Complete Ablation | 0
  Incomplete Ablation | 3

ADVERSE EVENTS:
Time Frame: up to 16 months
Description: Serious adverse effects" (SAE) are defined as pneumothorax requiring chest tube, bleeding requiring balloon tamponade or leading to respiratory failure, hypoxemia (SpaO2 <90% for > 1 min) during bronchoscopy, post-bronchoscopy pneumonitis with need of supplemental oxygen.
Arm/Group | Bronchoscopic Laser Ablation, Cone-beam CT(CBCT)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bronchoscopic Laser Ablation, Cone-beam CT(CBCT) (N=4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03707925/Prot_SAP_000.pdf